CLINICAL TRIAL: NCT05008757
Title: Comparison of Indirect Calorimetry by Q-NRG With Deltatrac II in Healthy Volunteers
Brief Title: Comparison of Indirect Calorimetry by Q-NRG With Deltatrac II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, University of Liege
Other Study IDs: B7072021000024
Record Dates: First submitted 2021-07-09; First posted 2021-08-17 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Indirect Calorimetry
Keywords: indirect calorimetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no drug — no intervention

SUMMARY:
Comparison of indirect calorimetry by Q-NRG (Cosmed) with Deltatrac II (Datex)

DETAILED DESCRIPTION:
The aim of the present study is to compare the measured resting energy expenditure by Q-NRG (Cosmed) with Deltatrac II (Datex), in healthy volunteers.

Q-NRG is a new device. It is relevant to compare its results with the blog standard calorimeter, the Deltratrac II.

The study will include sports healthy subjects. The could benefit from the determination of their resting energy expenditure in order to adapt their nutritional intakes.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult
* sport practice > 1h per day at moderate intensity

Exclusion Criteria:

* refusal to participate
* unable to give a consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers who practice more than 1 hour per day at moderate intensity
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
resting energy expenditure | during the calorimetry
  comparison of resting energy expenditure measured using Q-NRG calorimeter with resting energy expenditure measured using Deltatrac II

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Rousseau, MD, PhD, Principal Investigator — University Hospital of Liège, Belgium
Locations (1):
- Marjorie Fadeur, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No